CLINICAL TRIAL: NCT04789447
Title: Comparison of Initial CT Findings and CO-RADS Stage in COVID-19 Patients With PCR, Inflammation and Coagulation Parameters in Diagnostic and Prognostic Perspectives
Brief Title: Initial CT Findings and CO-RADS Stage in COVID-19
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: CT-19
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Covid19; SARS-CoV Infection; Pneumonia, Viral
Keywords: COVID-19; SARS-CoV2 RT-PCR Testing; Thorax; Computerized Tomography; Mortality; Prognosis
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients in hospital: All patients aged 18 years and over, positive for SARS-CoV-2 PCR test and / or Covid-19 treatment with signs of Covid-19 disease on CT

SUMMARY:
This study aims to determine whether patients with different real-time reverse transcriptase-polymerase chain reaction (PCR), chest computed tomography (CT) and laboratory findings have different clinical outcomes.

DETAILED DESCRIPTION:
This study aims to determine the rates of PCR positivity and CT findings in hospitalized patients with a diagnosis of COVID-19, to determine whether there is a difference in mortality and need for ICU between patients grouped according to the PCR positivity and presence of CT findings, and to evaluate the effect of the CO-RADS stage on these outcomes. Moreover, it is to compare the effects of inflammation and coagulation markers and CO-RADS stage on the severity of the disease

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over,
* Having SARS-CoV-2 RT-PCR test and chest CT examinations performed at the time of application or within 24 hours after admission
* RT-PCR positivity in nasopharyngeal swabs sample, and/or the presence of clinical and laboratory findings of SARS-CoV-2 infection and/or the presence of COVID-19-compatible radiological findings in chest CT, and being diagnosed with COVID-19

Exclusion Criteria:

* Patients with negative SARS-CoV-2 PCR test, pneumonia on CT but not given Covid-19 treatment by not considering Covid-19 by their doctor will not be included.
* Patients whose data are not available
* Patients with poor CT image quality
* Patients who were transferred to another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with Covid-19 in a two tertier hospital in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 895 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
mortality | up to 30 days
  mortality during hospitalization and within 14 days after hospitalization

SECONDARY OUTCOMES:
need for intensive care | up to 30 days
  need for intensive care during hospitalization and within 30 days after hospitalization
need for intenvasive mechanical ventilation | up to 30 days
  need for intenvasive mechanical ventilation during hospitalization and within 30 days after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Han Training and Rsearch Hospital
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided